CLINICAL TRIAL: NCT05823857
Title: Effect of Aquatic Exercise on Paraspinal and Gluteal Morphology and Function in Patients With Chronic Low Back Pain
Brief Title: Effect of an Aquatic Exercise Program in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Maryse Fortin, PhD, CAT(C), Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCER-21-22-35
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-11

CONDITIONS: Chronic Low-back Pain; Muscle Atrophy; Diagnostic Imaging; Exercise Therapy
Keywords: low back pain; musculoskeletal rehabilitation; aquatic therapy; standard care; diagnostic imaging; muscle morphology; randomized controlled trial
MeSH Terms: conditions — Muscular Atrophy; Low Back Pain | interventions — Aquatic Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: Pilot randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aquatic Therapy (Experimental): Aquatic exercise program including trunk stabilization, upper body, lower body strengthening and flexibility exercises and aerobic conditioning. Supervised 10-week program, 2 times a week.
  Interventions: Other: Aquatic Therapy
- Standard Care (Experimental): Standard care program including strengthening, flexibility, aerobic conditioning, modalities and manual mobilization techniques. Supervised 10-week program, 2 times a week.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Aquatic Therapy — Participants in this experimental intervention group will perform trunk stabilization, which will be based on a variety of aquatic exercises in different positions, intended to activate the multifidus and transverse abdominis in a co-contraction. Additionally, hip exercises will be completed to promote the strengthening of the gluteus maximus, gluteus medius, and gluteus minimus muscles. The aim of these exercises is to enhance the strength and dynamic stability of the spine and its surrounding musculature in a functional and yet non-weight-bearing way. Each exercise will be performed 10 times while sustaining the muscles co-contraction for 5-10 seconds and will be progressed gradually. Each training session (60 minutes) will be supervised by a Certified Athletic Therapist and take place in the PERFORM AT Clinic/Swim Ex pool.
  Arms: Aquatic Therapy
Other: Standard Care — Participants in this experimental intervention group will receive the standard LBP treatment in the PERFORM Athletic Therapy clinic.Two Certified Athletic Therapists (AT) will be conducting the sessions. The ATs will complete a thorough assessment of the eligible participants with chronic LBP and administer a range of interventions including stretching, strengthening and stabilization exercise, aerobic conditioning, and manual mobilization techniques. Other modalities could include application of ice and heat, ultrasound, and transcutaneous electrical nerve stimulation (TENS).
  Arms: Standard Care

SUMMARY:
The goal of this pilot randomized controlled trial is to compare the effects of aquatic therapy versus standard care on paraspinal and gluteal morphology and function in individuals with chronic low back pain.The main questions it aims to answer are:

1. What are the effects of aquatic therapy versus standard care on a) paraspinal and gluteal muscle size, composition (e.g., fatty infiltration) and b) lumbar and gluteal muscle strength in individuals with chronic LBP?
2. Is aquatic therapy more effective than standard care to improve pain, function and psychological factors (e.g., kinesiophobia, catastrophizing, anxiety, and depression)?
3. Is using a digital application "play the pain" feasible to monitor pain levels and the activities that participants used to cope with pain?

Participants will be assigned to either the aquatic therapy group or standard care group where they will undergo a 10-week intervention including two 60-minute session per week.

ELIGIBILITY:
Inclusion Criteria:

1. chronic nonspecific LBP (>3 months), defined as pain in the region between the lower ribs and gluteal folds, with or without leg pain
2. currently seeking care for LBP
3. aged between 18 and 65 years old
4. English or French speakers
5. have a score of "moderate" or "severe" disability on the modified Oswestry Low Back Questionnaire
6. do not currently engaged in sports or fitness training specifically for the lower back muscles (3 months prior the beginning of the trial).

Exclusion Criteria:

1. evidence of nerve root compression or reflex motor signs deficits
2. previous spinal surgery or vertebral fractures
3. other major lumbar spine structural abnormalities
4. comorbid health conditions that would prevent active participation in exercise programs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Change in multifidus muscle size (cross-sectional area) in cm^2 | Baseline, 10-week
  Multifidus muscle cross-sectional area measurements will be obtained from magnetic resonance imaging (MRI).
Change in gluteal muscle size (cross-sectional area) in cm^2 | Baseline, 10-week
  Gluteal muscle cross-sectional area measurements will be obtained from magnetic resonance imaging (MRI).
Percent change in multifidus muscle fatty infiltration in | Baseline, 10-week
  Multifidus muscle fatty infiltration (composition) measurements will be obtained from magnetic resonance imaging (MRI).
Percent change in gluteal muscle fatty infiltration | Baseline, 10-week
  Gluteal muscle fatty infiltration (composition) measurements will be obtained from magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Point score change in12-item Short Form Health Survey (SF-12) | Baseline, 10-week
  The 12-item Short Form Health Survey (SF-12) is the condensed form of the previous 36-item SF-12 Survey. The SF-12 is used to assess health-related quality of life. The 12-item survey consists of 8 domains that assess both physical and mental health composite scores (PCS and MCS). While the SF-12 is weighted and summed to provide a score for both the PCS and MCS. The score of the 12 questions can range from 0 (worst level of health) to 100 (highest level of health).
Point score change in Oswestry Low Back Pain Disability Index (ODI) score | Baseline, 10-week
  The ODI is used to measure the patient's level of disability in relation to LBP. It is a 10-item scale where each item is rated from 0-6. Higher scores are indicative of greater disability.
Point score change in Tampa Scale of Kinesiophobia (TSK) | Baseline, 10-week
  The TSK measures pain-related fear in an individual through a 13-item scale. The scores range between 17 and 68 with increasing scores indicating a greater level of kinesiophobia.
Point score change in The Pain Catastrophizing Scale (PCS) | Baseline, 10-week
  The PCS is a 13-item questionnaire that assesses an individual's level of catastrophizing. Each item is rated from 0-4 for a possible total of 52. Higher scores are indicative of a greater level of catastrophizing.
Point score change in The Hospital Anxiety and Depression Scale (HADS) | Baseline, 10-week
  The HADS is a 14-item questionnaire used to assess a patient's level of depression and anxiety. Each item is rated from 0-3 with either depression or anxiety having scores between 0 and 21. Higher scores are indicative of greater levels of anxiety and depression.
Point score change in Insomnia Severity Index (ISI) | Baseline, 10-week
  The ISI is a 7-item questionnaire used to assess sleep disturbances. Each item is rated from 0 to 4 and the total score is added. Higher scores are indicative of greater sleep disturbances.
Point score change in The International Physical Activity Questionnaire (IPAQ) | Baseline, 10-week
  The IPAQ is a self-reported log of metabolic equivalent (MET)-minutes per week. The level of physical activity is rated either vigorous, moderate, walking and sitting and must be assigned to the right category. The number of minutes per category is then added up and assessed.
Point score change in Visual Numerical pain rating scale (NPR) | Baseline, 10-week
  The NPR for pain is a rating system from 0 to 10 with 0 being no pain and 10 worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Maryse Fortin, PhD, Principal Investigator — Concordia University, Montreal
Locations (1):
- PERFORM Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaillancourt N, Montpetit C, Rosenstein B, Fortin M. Aquatic therapy compared to standard care for chronic low back pain: a randomized controlled trial. Pain Manag. 2026 Jan 13:1-13. doi: 10.1080/17581869.2026.2613633. Online ahead of print. PMID 41527881
- [Derived] Rosenstein B, Montpetit C, Vaillancourt N, Dover G, Khalini-Mahani N, Weiss C, Papula LA, Melek A, Fortin M. Effect of aquatic exercise versus standard care on paraspinal and gluteal muscles morphology in individuals with chronic low back pain: a randomized controlled trial protocol. BMC Musculoskelet Disord. 2023 Dec 18;24(1):977. doi: 10.1186/s12891-023-07034-0. PMID 38110922